CLINICAL TRIAL: NCT02850458
Title: Clinical Results of Implant-retained Mandibular Overdentures in Edentulous Patients: A 5-year Retrospective Study
Brief Title: Clinical Results of Implant-retained Mandibular Overdentures in Edentulous Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ji-hua Chen (Other)
Responsible Party: Sponsor-Investigator, Ji-hua Chen, Professor and Dean of the Department of Prosthodontics, School of Stomatology, Fourth Military Medical University, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Other Study IDs: IRB-REV-2016036
Record Dates: First submitted 2016-07-25; First posted 2016-08-01 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- implant retained-overdentures with the attachment of bar: patients treated with implant-retained overdentures,and the attachment is bar
  Interventions: Device: implant-retained overdentures
- implant retained-overdentures with the attachment of magnet: patients treated with implant-retained overdentures,and the attachment is magnet
  Interventions: Device: implant-retained overdentures

INTERVENTIONS:
Device: implant-retained overdentures — patients treated with an implant-retained overdenture in the mandible

SUMMARY:
The purpose of this study is to evaluate the clinical results of implant-retained mandibular overdentures in edentulous patients.

DETAILED DESCRIPTION:
The survival of implants,condition of the peri-implant soft tissue were evaluated. And patients' perceptions regarding the outcome were assessed on visual analog scales (VAS), oral health impact profile-14 (OHIP) and semantic differential scale questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated with implant retained overdentures
2. With the ability to read and sign the informed consent document

Exclusion Criteria:

1. Jaw radiotherapy treatment before and after implanting
2. Patients who suffered with mental and psychological disease will influence their oral health normal maintenance
3. Can not read and sign the informed consent document

Ages: 45 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated with implant retained overdentures at the Department of Prosthodontics, School of Stomatology of the Fourth Military Medical University between July 2011 to May 2014.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Survival of implants | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Gingival Bleeding on Probing | through study completion, an average of 1 year
  Gingival bleeding on probing (BOP) using the modified sulcus bleeding index for implants. Scale equals 0 = No bleeding when periodontal probe is passed along the gingival margin;1 = Isolated bleeding spots visible;2 = Blood forms a confluent red line on the gingival margin;3 = Heavy or profuse bleeding
Pocket depths | through study completion, an average of 1 year
  Pocket depths measured around implants in millimeter (mm)
Marginal bone loss | through study completion, an average of 1 year

OTHER OUTCOMES:
patients' satisfaction | through study completion, an average of 1 year
  patients' satisfaction were assessed on visual analog scales (VAS)
oral health-related quality of life | through study completion, an average of 1 year
  Patients completed a 14-item Oral Health Impact Profile (OHIP-14) to assess oral health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yong jin chen, Principal Investigator — IRB of Stomatological Hospital of FMMU,PLA
Locations (1):
- Stomatological Hospital of Fourth Military Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes